CLINICAL TRIAL: NCT05268575
Title: Comparative Study on Endoscopic Treatments for Hemorrhoids (METHOD): a Multicenter, Randomized Controlled Clinical Trial
Brief Title: A Study on the Endoscopic Treatments of Hemorrhoids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fangyu Wang (Other)
Collaborators: The Second Affiliated Hospital of Nanjing University of Chinese Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Fangyu Wang, Professor Wang, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZQH-KYLLSL-21-15
Record Dates: First submitted 2022-02-10; First posted 2022-03-07 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Pharmaceutical Preparations; Equipment and Supplies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- endoscopic sclerotherapy (Experimental): Patients with hemorrhoids will be treated with endoscopic sclerotherapy. Injection site is submucosa of hemorrhoid nucleus. Sclerosing agent makes the submucosal tissue fibrotic, and then fixes the hemorrhoidal tissue.
  Interventions: Other: performing endoscopy
- endoscopic rubber band ligation (Experimental): Patients with hemorrhoids will be treated with endoscopic rubber band ligation. The ligature position is above the mucosa of the hemorrhoid nucleus. Ligation of hemorrhoidal tissue can lead to ischemic necrosis of the prolapsed mucosa, which in turn leads to scar fixation. At the same time, the ligature also has the effect of lifting the tissue upward.
  Interventions: Other: performing endoscopy
- endoscopic sclerotherapy combined with rubber band ligation (Experimental): Patients with hemorrhoids will be treated with endoscopic sclerotherapy combined with rubber band ligation. Sclerotherapy first, followed by rubber band ligation. Sclerotherapy injection reduces the likelihood of ligature dislodgement.
  Interventions: Other: performing endoscopy

INTERVENTIONS:
Other: performing endoscopy — Hemorrhoids will be treated by endoscopic sclerotherapy or endoscopic rubber band ligation or endoscopic sclerotherapy combined with rubber band ligation
  Other Names: drugs; device

SUMMARY:
Hemorrhoids is one of the most common anorectal diseases, can occur at any age and gender. Hemorrhoids generally do not have very serious clinical manifestations, but often bring huge life pressure and psychological burden to patients, so effective treatment is necessary. Traditional surgical treatment techniques, such as hemorrhoidectomy, may have defects such as anal pain and long recovery time. Recently, endoscopic hemorrhoid treatment has become a safe, effective and rapid rehabilitation treatment. Treatment of hemorrhoids treatment including endoscopic sclerotherapy, endoscopic rubber band ligation, endoscopic sclerotherapy combined with rubber band ligation, the three kinds of treatment methods have their own advantages, but existing research at home and abroad is still less and the comparison of various treatment methods lack of consensus. Our study is to compare the three kinds of treatment methods.

DETAILED DESCRIPTION:
In this trial, investigators plan to conduct a multicenter, randomized controlled clinical trial. The leader of the sponsoring organization strictly implements oversight of the protocol. Investigators intend to compare the total efficiency of the endoscopic sclerotherapy group, the endoscopic rubber band ligation group, and the endoscopic sclerotherapy combined with rubber band ligation group for the treatment of hemorrhoids. The Department of Gastroenterology at Jinling Hospital will take full charge of this trial, including recruitment of patients, endoscopic treatment, in-hospital nursing, follow-up work, etc. Informed consent forms from every patient will be signed before enrollment, and approval from the Ethical Committees of Jinling Hospital has been obtained.

After patients will be admitted to the hospital and sign informed consent, they will be randomly assigned to the endoscopic sclerotherapy group, the endoscopic rubber band ligation group, and the endoscopic sclerotherapy combined with rubber band ligation group in a 1:1:1 ratio of 130 patients in each group, and the assignment will be done by a mobile client randomization tool. Patients in each group completed bowel preparation according to the same requirements and performed the appropriate endoscopic treatment. The sclerosing agent is polydocanol and the ligature model is MBL-6-F.

Our main observation is the overall effectiveness rate (the ratio of the number of people whose symptoms improved and the number of people whose symptoms completely disappeared to the total number of people). Our secondary observation indicators are the incidence of complications (such as urinary retention, prostatic abscess, fecal incontinence, rectal stricture, infection, bacteraemia, etc.) within 1 year after hemorrhoid treatment, the presence of new symptoms within 1 year after treatment, the recurrence rate after treatment, patient satisfaction, endoscopic performance of hemorrhoids, intraoperative conditions, hospital days, hospital costs, the need for retreatment due to recurrence or worsening of symptoms, blood routine, urine routine, fecal routine, coagulation function, blood biochemistry, etc.

Investigators will observe the status of patients 48 hours after treatment, 3 month after treatment, 6 months after treatment, 9 months after treatment, and 1 year after treatment. Follow-up will be conducted through online questionnaires or telephone callbacks.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form.
2. Age 18-80 years with clinical symptoms of hemorrhoids.
3. Subjects able to follow the follow-up schedule, able to describe symptoms objectively and able to cooperate in completing the scale.
4. non-breastfeeding pregnant women and those with no pregnancy planned during the trial
5. not participating in various clinical trials in the 3 months prior to and during the trial
6. Not taking long-term anticoagulant drugs (e.g., clopidogrel, aspirin, triptans, etc.) or have stopped taking them for 5-7 days.

Exclusion Criteria:

1. those with severe organ insufficiency of the heart, brain, lungs and kidneys
2. those who cannot tolerate endoscopic treatment
3. those with severe coagulation disorders
4. men with a history of severe prostate enlargement
5. with severe intestinal diseases: colon malignancy, ulcerative colitis, Crohn's disease, anal fistula, anal fissure, acute thrombosed internal hemorrhoids
6. those who are allergic to sclerosing agents
7. Those who, in the opinion of the investigator, cannot be enrolled for any reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Total effective rate | one year
  Total effective rate includes effective rate and cure rate. Effective rate means that symptoms are better than before treatment；Cure rate refers to the percentage of symptoms that completely disappear.

SECONDARY OUTCOMES:
Incidence of complications | 1 year
  Incidence of complications such as urinary retention, anal stricture, etc. within 1 year
Incidence of new symptoms | 1 year
  Incidence of new symptoms such as bleeding, pain, etc. within 1 year
Recurrence rate after treatment | 1 year
  Recurrence rate after 1 year of treatment
Patient satisfaction | 1 year
  A questionnaire was used to obtain patients' responses regarding their satisfaction with the treatment, with the following three options: satisfied, indifferent, and dissatisfied.
Endoscopic presentation of hemorrhoids | 1 year
  Circumferential distribution of hemorrhoids, the diameter of the largest hemorrhoids, presence of red color signs (change in the color of the surface of the rectal column in accordance with the general rules for endoscopic findings of esophagogastric varices)
Intraoperative situation | 1 year
  The amount of intraoperative bleeding and whether the patient had discomfort during the operation.
Number of days in hospital | 1 year
  Number of days in hospital
Hospitalization Costs | 1 year
  Hospitalization Costs
Incidence of needing re-treatment | 1 year
  Need for retreatment due to recurrence or worsening of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamana T. Japanese Practice Guidelines for Anal Disorders I. Hemorrhoids. J Anus Rectum Colon. 2018 May 25;1(3):89-99. doi: 10.23922/jarc.2017-018. eCollection 2017. PMID 31583307
- [Background] Madoff RD, Fleshman JW; Clinical Practice Committee, American Gastroenterological Association. American Gastroenterological Association technical review on the diagnosis and treatment of hemorrhoids. Gastroenterology. 2004 May;126(5):1463-73. doi: 10.1053/j.gastro.2004.03.008. No abstract available. PMID 15131807
- [Background] Ma W, Guo J, Yang F, Dietrich CF, Sun S. Progress in Endoscopic Treatment of Hemorrhoids. J Transl Int Med. 2020 Dec 31;8(4):237-244. doi: 10.2478/jtim-2020-0036. eCollection 2020 Dec. PMID 33511050
- [Background] Davis BR, Lee-Kong SA, Migaly J, Feingold DL, Steele SR. The American Society of Colon and Rectal Surgeons Clinical Practice Guidelines for the Management of Hemorrhoids. Dis Colon Rectum. 2018 Mar;61(3):284-292. doi: 10.1097/DCR.0000000000001030. No abstract available. PMID 29420423
- [Background] Awad AE, Soliman HH, Saif SA, Darwish AM, Mosaad S, Elfert AA. A prospective randomised comparative study of endoscopic band ligation versus injection sclerotherapy of bleeding internal haemorrhoids in patients with liver cirrhosis. Arab J Gastroenterol. 2012 Jun;13(2):77-81. doi: 10.1016/j.ajg.2012.03.008. Epub 2012 Apr 24. PMID 22980596
- [Background] Kanellos I, Goulimaris I, Christoforidis E, Kelpis T, Betsis D. A comparison of the simultaneous application of sclerotherapy and rubber band ligation, with sclerotherapy and rubber band ligation applied separately, for the treatment of haemorrhoids: a prospective randomized trial. Colorectal Dis. 2003 Mar;5(2):133-8. doi: 10.1046/j.1463-1318.2003.00395.x. PMID 12780901
- [Background] Abiodun AA, Alatise OI, Okereke CE, Adesunkanmi AK, Eletta EA, Gomna A. Comparative study of endoscopic band ligation versus injection sclerotherapy with 50% dextrose in water, in symptomatic internal haemorrhoids. Niger Postgrad Med J. 2020 Jan-Mar;27(1):13-20. doi: 10.4103/npmj.npmj_128_19. PMID 32003357